CLINICAL TRIAL: NCT06995365
Title: Patient-centered Precision Medicine Lab Result Communication for Older Adults - Validation and Refinement of an Existing Chronic Kidney Disease (CKD) Risk Model
Brief Title: Refining Risk Prediction Models for Older Adults Using Electronic Health Records
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Associate Professor of Medicine, University of California, Los Angeles
Other Study IDs: IRB-25-0471
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Predictive Modeling
Keywords: Lab Result Communication; Risk Stratification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Risk Prediction Model — This study analyzes retrospective electronic health record (EHR) data from older adults to refine and validate a predictive model for other conditions in future studies.

SUMMARY:
This study aims to improve how lab results are communicated to older adults by refining a predictive model that uses electronic health record (EHR) data. The model was originally developed to estimate the risk of chronic kidney disease (CKD) progression. Researchers will use existing health data to test and improve the accuracy of the model and explore how it might be adapted for use in other health conditions. The study does not involve direct interaction with patients and is conducted entirely using de-identified data in a secure environment.

ELIGIBILITY:
Inclusion Criteria include, but are not limited to:

* being over the age of 65; having at least 5 years of clinical follow up; and having a serum creatinine lab test conducted

Exclusion Criteria:

* Patients younger than 65 years old
* Patients with less than 5 years of clinical follow-up
* Patients from health systems outside of the UC Health network.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 65 and older who received care within the UCLA or UC Health system, have at least 5 years of clinical follow-up, and have had a serum creatinine test. Data are drawn from existing electronic health records.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Performance of the Risk Prediction Model | Up to 5 years of retrospective follow up
  Evaluate the predictive performance of a machine learning-based risk model using retrospective Electronic Health Records (EHR) data. The model estimates the likelihood of disease progression in older adults. The model should be designed to be adaptable to various clinical conditions. Metrics include Area Under the Receiver Operating Characteristic Curve (AUC-ROC), sensitivity, and specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Health System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No